CLINICAL TRIAL: NCT01872468
Title: Effectiveness of an Structured Intervention in Patients With Chronic Kidney Failure to Reduce the Progression of the Illness.
Brief Title: Effectiveness of a Structured Intervention to Reduce the Progression of Chronic Kidney (RENAP Study)
Acronym: RENAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gerencia de Atención Primaria, Madrid (Other Government)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Marta Sanchez-Celaya del Pozo, Phycisian doctor, Gerencia de Atención Primaria, Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 09/90845
Record Dates: First submitted 2013-06-03; First posted 2013-06-07 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Renal Insufficiency Chronic
Keywords: Glomerular filtration Rate.; Primary Health Care.; Cluster Clinical Trial.
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): There is not intervention in this group.
- Structured intervention (Active Comparator): Initial training session based on significant learning and follow up visits every four months at physicians and nurses´ offices over a two-year period
  Interventions: Behavioral: Structured intervention

INTERVENTIONS:
Behavioral: Structured intervention — Initial training session based on patient personal experiences and reflexion (30 minutes). CKD learning session (30 minutes). Personal plan of actions to cope with own disease (30 minutes. Discussion of doubts (30 minutes). Follow up visits every four months at physicians and nurses´ offices over a two-year period
  Arms: Structured intervention

SUMMARY:
The propose of study is to study if an informative intervention and a structured follow-up carried out in health centres of primary care in patients with chronic kidney failure, stage 3, is more effective than the current follow-up in slowing the disease progression measured by the glomerular filtration rate.

DETAILED DESCRIPTION:
Main objective: To study if an informative intervention and a structured follow-up carried out in health centres of primary care in patients with chronic kidney failure, stages 3, is more effective than the current follow-up in slowing the disease progression measured by the glomerular filtration rate .

Secondary objectives: Determining the effectiveness of the intervention to improve the blood pressure control of the patients with chronic kidney failure and to improve the degree of control of the glucose levels and glycosylated haemoglobin of the diabetic patients with chronic kidney failure.

Design: A clinical trial controlled with a random assignment by conglomerates with parallel groups.

Setting: Multi-centre study in Primary Care Health Centres(Madrid Health Service).

Subjects of the study: 540 patients over 18 years old, diagnosed of light-moderate chronic kidney failure that consent to participate.

Data collection: The variable of the main answer will be the creatinine clearance measured in ml/min. Demographic variables of morbidity and prognosis: clinical, analytical, anthropometrical, adherence to processing and consumption of medicines will be collected.

Intervention: Initial educational session based on the significant learning and quarterly follow-up in surgery of medicine and nursing for 2 years.

Analysis: By intention of treating. Descriptive statistics of each variable and statistical analytical univariate and multivariate (multiple linear regression) will be carried out. The explanatory variable in the analysis multivariate will be the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Willing and able to give informed consent for participation in the study.
* Ability to understand study procedures and to comply with them for the entire length of the study.
* Registered episode on electronic medical records in Primary Care with the diagnosis of Chronic Kidney Disease (CKD) stage 3 or confirmation of CKD by a second blood sample in risk patients with suspected CKD( owing to a blood sample taken at least three months before

Exclusion Criteria:

* Inability or unwillingness to give written informed consent.
* Severe psychiatric conditions including depression and major affective disorders registered on medical records.
* Disabled and unable to attend Health Centre.
* Severe CKD, defined as glomerular filtration rate (GFR) < 30 ml/min/1,73m2.
* Patients undergoing dialysis or kidney transplantation.
* Patients hemodynamically unstable with impaired kidney function (Eg. Cardiac Failure, unstable angina pectoris).
* Acute kidney failure.
* Patients with an episode of impaired kidney perfusion on the last month (Eg. Severe hemorrhage, burns, dehydration, major trauma).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2011-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Creatinine clearance | 2 years
  Glomerular filtration rate measured by Modification of Diet in Renal Disease (MDRD)formula and expressed in ml/min. The MDRD formula estimates the glomerular filtrate through the levels of creatinine plasma, sex and age.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Sánchez-Celaya, Doctor, Principal Investigator — Gerencia Atención Primaria. Madrid
Locations (1):
- Gerencia Atencion Primaria, Madrid, Madrid, Spain